CLINICAL TRIAL: NCT06829342
Title: The Role of Sensory Deficits in the Neural Control of Balance During Walking in Parkinson's Disease
Brief Title: Stochastic Resonance Stimulation Effect on Gait Stability in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Parkinson's Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1759595-5
Record Dates: First submitted 2025-02-03; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stochastic Resonance (SR) (Experimental): During this condition, participants will walk on the treadmill while receiving SR stimulation at their individual optimal intensity (SR) with and without visual perturbations.
  Interventions: Device: Stochastic Resonance (SR)
- No Stochastic Resonance (no-SR) (No Intervention): During this condition, participants will walk on the treadmill while receiving no SR stimulation (no-SR) with and without visual perturbations.

INTERVENTIONS:
Device: Stochastic Resonance (SR) — The system consists of six linear isolated stimulators (STMISOLA, Biopac Systems, Inc., Goleta, USA). The SR signal (Gaussian White Noise, zero mean) will be generated through a 16 bit PCI 6733 National Instruments multifunction data acquisition card by a custom LabView program. The stimulation sites include the ankle, lateral soleus, peroneus longus, and tibialis anterior muscles and the hip.
  Arms: Stochastic Resonance (SR)

SUMMARY:
The present study explored the use of a technique called stochastic resonance (SR) stimulation that may help individuals with Parkinson Disease maintain balance while walking on challenging surfaces. Impaired balance represents one of the disease symptoms, putting people at risk for falls, partly due to impaired processing of sensory information. SR uses light electrical signals to improve the way the body detects sensations. We wanted to test if SR could help people with Parkinson disease stay steadier while walking. Each participant's optimal SR intensity was determined before they walked on a treadmill in a virtual environment that created visual disturbances to challenge their balance. We measured how much their body swayed, how they placed their feet, and how their ankles moved during the walking tasks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson Disease
* Hoehn and Yahr (H&Y) stage ≤ III
* Can walk independently for at least 2 minutes without an assistive device or orthosis
* Ability to communicate discomfort during testing
* Can follow multi-step commands
* Scored at least 24/30 on the Montreal Cognitive assessment (MoCA)

Exclusion Criteria:

* Any head, neck, or face injury in the six months prior to the study (e.g., concussion, eye injury)
* History of vestibular or ocular dysfunction
* Currently taking any medications affecting balance (i.e. antibiotics)
* Injuries to lower extremities affecting balance in the past six months
* Pregnancy
* Any neurological disorders other than Parkinson's disease (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 minutes, CNS neoplasm, history of stroke)
* Unstable cardiac or pulmonary disease
* Clinically obese (BMI 30 or above)
* Any metal implant in the feet or legs that is close to the stimulating electrodes
* A known allergy to medical-grade adhesives
* Any other comorbidity affecting the ability to safely walk without assistance for at least 2 minutes
* Exhibited severe dyskinesia
* Did not respond to L-DOPA or other dopaminergic treatment
* Exhibited cardiovascular-autonomic or multiple-system symptoms indicative of a "Parkinsonism-plus" presentation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Change in the Center of Mass (CoM) excursion | Through study completion, an average of 1 year.
  For the visual perturbation trials, we will use CoM excursion as the primary outcome measure since it has been used in prior studies in children and adults using visual perturbation protocols. This is determined by comparing the average CoM during perturbed steps to non-perturbed steps for each participant, integrated across the first eight steps initiated by the heel strike that triggered the stimulus. We will measure CoM using kinetics and kinematic computed through a motion capture system(Qualysis).
  For the unperturbed trials, we will use margin of stability (MoS) as the primary outcome measure. MOS refers to the distance between extrapolated center of mass, which includes center of mass position and velocity, and the base of support. It has been previously used to measure balance in children with cerebral palsy and Parkinson Disease.

CONTACTS AND LOCATIONS:
Overall Officials: John J Jeka, PhD, Study Director — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided